CLINICAL TRIAL: NCT00035412
Title: St. John's Wort Versus Placebo in Social Phobia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R21AT000502-01A1 (NIH)
Record Dates: First submitted 2002-05-03; First posted 2002-05-06 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-07

CONDITIONS: Phobic Disorders
Keywords: Social phobia; Social anxiety; Anxiety; St. John' Wort; Wisconsin; Psychiatric; Mental health
MeSH Terms: conditions — Phobic Disorders; Phobia, Social; Anxiety Disorders; Psychological Well-Being | interventions — Hypericum extract LI 160

INTERVENTIONS:
Drug: St. John's Wort

SUMMARY:
The purpose of this study is to determine the effectiveness of St. John's Wort as compared to placebo (an inactive substance) in the treatment of outpatients with social phobia.

DETAILED DESCRIPTION:
Social Phobia is a prevalent and debilitating condition, with a lifetime prevalence rate to be 13.3 percent. Socially phobic patients have been found to be functionally impaired in the areas of education, employment and social relationships, to have poorer quality of life, and increased suicidal ideation and psychiatric comorbidity. Double-blind studies have found benzodiazepines, selective and non-selective MAOI inhibitors, several SSRIs, and the anticonvulsants pregabalin and gabapentin to be effective. However, side effects with these compounds suggests the need for better tolerated compounds, e.g., in the paroxetine multi-center trial (the only drug with an FDA approved indication), 27 percent reported somnolence, 26 percent nausea, and 37 percent of males reported delayed ejaculation; 34 percent of patients discontinued the trial early. There has been considerable worldwide interest in St. John's Wort (SJW) (Hypericum perforatum) as a treatment of mild to moderate depression. There have been 23 randomized trials suggesting SJW is more effective than placebo for the treatment of outpatients with mild to moderate depression. SJW is very well tolerated with mild side effects observed in only 2.5 percent of cases in a large (3250 patients) drug monitoring study. Pharmacokinetic studies have found Hypericum to have affinity for serotonin, dopamine and GABA alpha and GABA beta receptors, each of which have been implicated in social phobia, thus there is a suggestion that SJW may be effective for this disorder.

This will be a 12-week, double blind, placebo-controlled trial, designed to generate effect size data that will be used to determine sample size needed to power a definitive study. Forty patients will be randomized to either SJW (LI 160) or matching placebo. This will be a flexible-dose design, starting at 300 mg tid to a maximum of 1800 mg total per day. An intent-to-treat analysis will be employed. Subjects will be evaluated weekly for two weeks, then bi-weekly thereafter. The primary outcome measure will be the change from baseline to endpoint on the Liebowitz Social Anxiety Scale.

ELIGIBILITY:
Inclusion Criteria:

* Female patients: at least 2 years post-menopausal, surgically sterile, or practicing a medically acceptable method of contraception.
* Meets DSM-IV criteria for Social Phobia, generalized subtype, lasting 12 months in duration (phone screening will determine)

Exclusion Criteria:

* Primary diagnosis of major depression, dysthymia, panic disorder, schizophrenia, schizo-affective disorder, bipolar disorder, or PTSD
* Substance abuse or dependence in the past 6 months
* Vascular dementia or primary degenerative dementia of the Alzheimer's type
* Treatment with MAOIs, TCAs, SSRIs, venlafaxine, nefazodone, remeron, citalopram, or bupropion within 14 days of first visit.
* Fluoxetine within 14 days of first visit.
* Failure to respond to at least two adequate antidepressant trials for social anxiety.
* Investigational drugs within 30 days of baseline
* Known allergy or hypersensitivity to St. John's Wort
* Currently in behavior therapy for Social Phobia

ALL INQUIRIES WILL UNDERGO A PHONE SCREENING TO DETERMINE WHETHER THEY MEET ELIGIBLITY REQUIREMENTS.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2001-12; Study Completion 2004-08

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Kobak, PhD, Principal Investigator — Dean Foundation for Health, Research and Analysis; Leslie Taylor, MD, Principal Investigator — Dean Foundation for Health, Research and Analysis
Locations (1):
- The Dean Foundation for Health, Research, and Education, Madison, Wisconsin, United States

REFERENCES:
- See also: A non-profit foundation located in Middleton, Wisconsin, conducting clinical trials of psychiatric and medical therapies. — http://www.dean.org